CLINICAL TRIAL: NCT03036969
Title: Emergency Processes in Clinical Structures - EPICS-8: Gründe für Die Inanspruchnahme Der Notaufnahme Durch Patienten Mit Blauer, grüner Oder Gelber Triagekategorie Und Ambulantem Behandlungsbedarf
Brief Title: EPICS-8: Reasons for Emergency Department Utilization by Patients With Non-urgent Conditions
Acronym: EPICS-8
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Zentralinstitut für die Kassenärztliche Versorgung in Deutschland (Unknown)
Responsible Party: Principal Investigator, Martin Moeckel, Univ.-Prov., Charite University, Berlin, Germany
Other Study IDs: EPICS-8
Record Dates: First submitted 2017-01-24; First posted 2017-01-31 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Non-urgent Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non-urgent emergencies: Outpatients in the Emergency Department with the MTS-Triage category blue, green or yellow

SUMMARY:
EPICS-8: Reasons for Emergency Department utilization by patients with non-urgent conditions:

Emergency Departments (EDs) are an important interface between primary and secondary health care sectors in Germany. The number of outpatient visits in the ED´s is still increasing. The reasons for ED utilization by patients with non-urgent conditions are nearly unknown in Germany and will be investigated in this project.

DETAILED DESCRIPTION:
EPICS-8: Reasons for Emergency Department utilization by patients with non-urgent conditions:

Emergency Departments (EDs) are an important interface between primary and the secondary health care system in Germany. The number of outpatient visits in the ED´s is still increasing. The reasons for ED utilization by patients with non-urgent conditions are nearly unknown in Germany and will be explored in this project.

EPICS-8 is a pilot study to establish a research structure for the linkage of ED-data with data of the primary health care sector. Data linkage will be conducted for patients with the Manchester Triage System categories blue, green and yellow. A secondary aim of the EPICS-8 study is to develop a valid questionnaire for the assessment of reasons for ED utilization by non-urgent patients.

Primary objective:

Establishing of a research structure for the linkage of inhospital-data with data from the primary health care System. Records of 5,000 patients who attended one of the two EDs at the Charité University Medicine Berlin will be linked to Primary health care data.

Secondary objectives:

1. Development and testing of a questionaire for the identification of reasons for emergency department utilization by patients with non-urgent conditions (n=100)
2. Characterization and quantification of non-urgent emergencies
3. Explorative analysis of patient pathways and influencing factors for ED-visits with non-urgent conditions.

ELIGIBILITY:
Eligibility criteria for record linkage:

* Age>= 18 years
* Outpatients
* MTS-Triage category blue, green or yellow
* Treatment in one of the two participating EDs

Eligibility criteria for questionnaire pretest:

Inclusion Criteria:

* Age>= 18 years
* Outpatients
* MTS-Triage category blue, green or yellow
* Treatment in one of the two participating EDs
* Eligibility to understand the study purposes and give written informed consent

Exclusion Criteria:

* Dementia
* no sufficient German language skills
* patients with legal representatives

Ages: 18 Years to 115 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult men and women who are discharged after emergency treatment (outpatients) with an initial Manchester Triage Category of blue, green or yellow.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients with linkable records | 05/2016 - 05/2018
  The Primary outcome will be the proportion of patients with successful record linkage.

SECONDARY OUTCOMES:
Valid Questionnaire | 05/2016 - 05/2017
  A patients questionnaire for the assessment of Emergency Department utilization by non-urgent patients will be developed. The outcome of this work package will be a valid patient questionnaire.
Demographic characteristics of non-urgent ED patients | During the study period
  Descriptive analysis of demographic characteristics of ED patients with non-urgent conditions
Clinical characteristics of non-urgent ED patients | During the study period
  Descriptive analysis of clinical characteristics of ED patients with non-urgent conditions
Patient pathways for ED-Visits | 10/2017 - 05/2018
  Explorative analysis of patient pathways for ED-visits with non-urgent conditions
Influencing factors for ED-Visits | 10/2017 - 05/2018
  Explorative analysis of influencing factors for ED-visits with non-urgent conditions

CONTACTS AND LOCATIONS:
Overall Officials: Martin Möckel, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin - Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No